CLINICAL TRIAL: NCT00153036
Title: ECASS III - European Cooperative Acute Stroke Study III: A Placebo Controlled Trial of Alteplase (Rt-PA) in Acute Ischemic Hemispheric Stroke Where Thrombolysis is Initiated Between 3 and 4 Hours 30 Minutes After Stroke Onset
Brief Title: Rt-PA in the Treatment of Acute Ischemic Stroke
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Purpose: Treatment
Other Study IDs: 135.312
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-04

CONDITIONS: Cerebrovascular Accident
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Drug: rt-PA 0.9 mg/kg verum or placebo Intravenous

SUMMARY:
To collect additional confirmatory data on alteplase(rt-PA) in the European setting and to demonstrate that the treatment of patients between 3 and 4.30 hours of onset of symptoms of acute ischemic stroke with rt-PA compared to placebo-treated patients will result in an improved clinical outcome without increase of fatality rate.

ELIGIBILITY:
Inclusion Criteria:

* Female or male inpatients
* Age: 18 - 80 years.
* Clinical diagnosis of ischemic stroke causing a measurable neurological deficit defined as impairment of language, motor function, cognition and/or gaze, vision or neglect. Ischemic stroke is defined as an event characterized by the sudden onset of an acute focal neurologic deficit presumed to be due to cerebral ischemia after CT scan excludes hemorrhage.
* Onset of symptoms between 3 and 4 hours prior to initiation of administration of study drug.
* Stroke symptoms are to be present for at least 30 minutes and have not significantly improved before treatment. Symptoms must be distinguishable from an episode of generalized ischemia (i.e. syncope), seizure, or migraine disorder.
* Patient is willing to participate voluntarily and to sign a written patient informed consent. Informed consent will be obtained from each patient or the subject's legally authorized representative or relatives, or deferred where applicable, according to the regulatory and legal requirements of the participating country.
* Patients who are unable to sign but who are able to understand the meaning of participation in the study may give an oral witnessed informed consent. These patients have to make clear undoubtfully that they are willing to participate voluntarily and must be able to understand an explanation of the contents of he information sheet.
* Willingness and ability to comply with the protocol.

Exclusion Criteria:

* Evidence of intracranial hemorrhage (ICH) on the CT-scan.
* Symptoms of ischaemic attack began more than 4 hours and 30 minutes prior to infusion start or when time of symptom onset is unknown.
* Minor neurological deficit or symptoms rapidly improving before start of infusion.
* Severe stroke as assessed clinically (e.g. NIHSS>25) and/or by appropriate imaging techniques.
* Epileptic seizure at onset of stroke
* Symptoms suggestive of subarachnoid haemorrhage, even if the CT-scan is normal.
* Administration of heparin within the previous 48 hours and a thromboplastin time exceeding the upper limit of normal for laboratory
* History of prior stroke and concomitant diabetes. * Prior stroke within the last 3 months
* Platelet below 100,000/mm3. * Systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg, or aggressive management (IV medication) necessary to reduce BP to these limits.
* Blood glucose <50 or > 400 mg/dl (< 2.77 or > 22.15 mmol / l). * Known haemorraghic diathesis
* Patients receiving oral anticoagulants. * Manifest or recent severe or dangerous bleeding
* Known history of or suspected intracranial haemorrhage
* Suspected subarachnoid haemorrhage or condition after subarachnoid haemorrhage from aneurysm
* History of central nervous system damage (i.e. neoplasm, aneurysm, intracranial or spinal surgery)
* Haemorrhagic retinopathy,e.g. in diabetes (vision disturbances may indicate haemorrhagic retinopathy)
* Recent (less than 10 days) traumatic external heart massage, obstetrical delivery, recent puncture of a non-compressible blood-vessel (e.g. subclavian or jugular vein puncture.
* bacterial endocarditis, pericarditis.* Acute pancreatitis
* Documented ulcerative gastrointestinal disease during the last 3 months, oesophageal varices, arterial- aneurysm, arterial/venous malformation
* Neoplasm with increased bleeding risk

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 821 (Actual)
Dates: Start 2003-04; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
modified Rankin scale (mRS) 0-1 (favourable outcome) at Day 90 | at day 90

SECONDARY OUTCOMES:
Global outcome of four neurologic and disability scores combined | at day 90

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (142):
- Austria (10):
  - 135.312.43004 Boehringer Ingelheim Investigational Site, Graz
  - 135.312.43007 Boehringer Ingelheim Investigational Site, Innsbruck
  - 135.312.43010 Boehringer Ingelheim Investigational Site, Klagenfurt
  - 135.312.43001 Boehringer Ingelheim Investigational Site, Linz
  - 135.312.43012 Boehringer Ingelheim Investigational Site, Linz
  - 135.312.43013 Boehringer Ingelheim Investigational Site, Linz
  - 135.312.43008 Boehringer Ingelheim Investigational Site, Ma.Gugging/Klosterneuburg
  - 135.312.43006 Boehringer Ingelheim Investigational Site, Salzburg
  - 135.312.43003 Boehringer Ingelheim Investigational Site, Sankt Pölten
  - 135.312.43002 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (7):
  - 135.312.32006 O.L. Vrouwziekenhuis, Aalst
  - 135.312.32002 Boehringer Ingelheim Investigational Site, Anderlecht
  - 135.312.32014 Boehringer Ingelheim Investigational Site, Antwerp
  - 135.312.32001 Boehringer Ingelheim Investigational Site, Bruges
  - 135.312.32016 Boehringer Ingelheim Investigational Site, Godinne
  - 135.312.32011 Boehringer Ingelheim Investigational Site, Kortrijk
  - 135.312.32005 Boehringer Ingelheim Investigational Site, Leuven
- Czechia (3):
  - 135.312.42001 Boehringer Ingelheim Investigational Site, Ostrava
  - 135.312.42004 Boehringer Ingelheim Investigational Site, Ostrava-Vitkovice
  - 135.312.42002 Boehringer Ingelheim Investigational Site, Prague
- Denmark (4):
  - 135.312.45005 Boehringer Ingelheim Investigational Site, Aalborg
  - 135.312.45002 Boehringer Ingelheim Investigational Site, Aarhus
  - 135.312.45001 Boehringer Ingelheim Investigational Site, Copenhagen NV
  - 135.312.45004 Boehringer Ingelheim Investigational Site, Glostrup Municipality
- Finland (3):
  - 135.312.35801 Boehringer Ingelheim Investigational Site, Helsinki
  - 135.312.35805 Boehringer Ingelheim Investigational Site, Kuopio
  - 135.312.35802 Boehringer Ingelheim Investigational Site, Turku
- France (24):
  - 135.312.33009 Boehringer Ingelheim Investigational Site, Auch
  - 135.312.33016 Boehringer Ingelheim Investigational Site, Besançon
  - 135.312.33013 Boehringer Ingelheim Investigational Site, Bordeaux
  - 135.312.33017 Boehringer Ingelheim Investigational Site, Bourg-en-Bresse
  - 135.312.33008 Boehringer Ingelheim Investigational Site, Dijon
  - 135.312.33014 Boehringer Ingelheim Investigational Site, Grenoble Cédex 9
  - 135.312.33015 Boehringer Ingelheim Investigational Site, Lille
  - 135.312.33019 Boehringer Ingelheim Investigational Site, Limoges
  - 135.312.33001 Boehringer Ingelheim Investigational Site, Lyon
  - 135.312.33024 Boehringer Ingelheim Investigational Site, Mantes-la-Jolie
  - 135.312.33021 Boehringer Ingelheim Investigational Site, Meaux
  - 135.312.33002 Boehringer Ingelheim Investigational Site, Montpellier
  - 135.312.33004 Boehringer Ingelheim Investigational Site, Nancy
  - 135.312.33003 Boehringer Ingelheim Investigational Site, Nice
  - 135.312.33006 Boehringer Ingelheim Investigational Site, Paris
  - 135.312.33007 Boehringer Ingelheim Investigational Site, Paris
  - 135.312.33020 Boehringer Ingelheim Investigational Site, Pau
  - 135.312.33018 Boehringer Ingelheim Investigational Site, Perpignan
  - 135.312.33023 Boehringer Ingelheim Investigational Site, Pontoise
  - 135.312.33010 Boehringer Ingelheim Investigational Site, Saint-Herblain
  - 135.312.33005 Boehringer Ingelheim Investigational Site, Toulouse
  - 135.312.33012 Boehringer Ingelheim Investigational Site, Toulouse
  - 135.312.33011 Boehringer Ingelheim Investigational Site, Tours
  - 135.312.33022 Boehringer Ingelheim Investigational Site, Versailles
- Germany (19):
  - 135.312.49031 Boehringer Ingelheim Investigational Site, Altenburg
  - 135.312.49011 Boehringer Ingelheim Investigational Site, Bamberg
  - 135.312.49037 Boehringer Ingelheim Investigational Site, Beeskow
  - 135.312.49017 Boehringer Ingelheim Investigational Site, Bochum
  - 135.312.49008 Boehringer Ingelheim Investigational Site, Cologne
  - 135.312.49038 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 135.312.49041 Boehringer Ingelheim Investigational Site, Hamburg
  - 135.312.49023 Boehringer Ingelheim Investigational Site, Hanover
  - 135.312.49001 Boehringer Ingelheim Investigational Site, Heidelberg
  - 135.312.49014 Boehringer Ingelheim Investigational Site, Leipzig
  - 135.312.49020 Boehringer Ingelheim Investigational Site, Ludwigshafen am Rhein
  - 135.312.49004 Boehringer Ingelheim Investigational Site, Magdeburg
  - 135.312.49003 Boehringer Ingelheim Investigational Site, Mainz
  - 135.312.49018 Boehringer Ingelheim Investigational Site, Mannheim
  - 135.312.49002 Boehringer Ingelheim Investigational Site, Minden
  - 135.312.49006 Boehringer Ingelheim Investigational Site, München
  - 135.312.49005 Boehringer Ingelheim Investigational Site, Siegen
  - 135.312.49025 Boehringer Ingelheim Investigational Site, Teupitz
  - 135.312.49009 Boehringer Ingelheim Investigational Site, Wiesbaden
- Greece (3):
  - 135.312.30004 Boehringer Ingelheim Investigational Site, Athens
  - 135.312.30005 Boehringer Ingelheim Investigational Site, Larissa
  - 135.312.30002 Boehringer Ingelheim Investigational Site, Thessaloniki
- Hungary (3):
  - 135.312.36002 University of Debrecen, Debrecen
  - 135.312.36001 Aladár Petz County Hospital, Győr
  - 135.312.36006 BAZ County and Teaching Hospital, Miskolc
- Italy (16):
  - 135.312.39020 Università degli Studi, Coppito (aq)
  - 135.312.39013 A. O. Universitaria di Careggi, Florence
  - 135.312.39019 Ospedale Santa Maria Annunziata, Florence
  - 135.312.39022 Ospedale di Imperia, Imperia
  - 135.312.39024 Istituto Scientifico San Raffaele, Milan
  - 135.312.39002 A. O. di Padova - Policlinico Universitario, Padua
  - 135.312.39005 A. O. di Perugia - Policlinico Monteluce, Perugia
  - 135.312.39023 P. O. di Piacenza, Piacenza
  - 135.312.39016 A. O. Ospedale Santa Corona, Pietra Ligure (sv)
  - 135.312.39006 Ospedale Santa Chiara, Pisa
  - 135.312.39003 A. O. Arcispedale "Santa Maria Nuova", Reggio Emilia
  - 135.312.39001 A. O. Policlinico Umberto I, Roma
  - 135.312.39025 Università di Roma "La Sapienza", Roma
  - 135.312.39018 Ospedale S. Maria della Misericordia, Udine
  - 135.312.39009 Ospedale Maggiore di BorgoTrento, Verona
  - 135.312.39004 Ospedale Civile, Vicenza
- Netherlands (2):
  - 135.312.31001, Amsterdam
  - 135.312.31007 Medisch Spectrum Twente, Enschede
- Norway (3):
  - 135.312.47001 Boehringer Ingelheim Investigational Site, Bergen
  - 135.312.47003 Boehringer Ingelheim Investigational Site, Trondheim
  - 135.312.47006 Boehringer Ingelheim Investigational Site, Tønsberg
- Poland (5):
  - 135.312.48004 Medical University of Gdansk, Gdansk
  - 135.312.48005 Dept. of Neurology, Regenerative and Cerebrovascular Disease, Katowice
  - 135.312.48006 Wojewodship Specialistic Neuropsychiatric Centre in Opole, Opole
  - 135.312.48001 Institute of Psychiatry & Neurology in Warsaw, Warsaw
  - 135.312.48002 Dr. Anna Gostynska Wolski Hospital, Warsaw
- Portugal (4):
  - 135.312.35101 Hospitais da Universidade de Coimbra, Coimbra
  - 135.312.35106 Hospital de Santa Maria, Lisbon
  - 135.312.35102 Hospital de Santo António, Porto
  - 135.312.35105 Hospital de São Sebastião, EPE, Santa Maria da Feira
- Slovakia (5):
  - 135.312.42103 NEURON PLUS s.r.o, Bratislava
  - 135.312.42102 Hospital Levoca, Levoča
  - 135.312.42104 Jessenius Faculty of Medicine Commenius University, Martin
  - 135.312.42101 Faculty Hospital, Nitra
  - 135.312.42105 Boehringer Ingelheim Investigational Site, Trnava
- Spain (13):
  - 135.312.34019 Boehringer Ingelheim Investigational Site, Albacete
  - 135.312.34006 Boehringer Ingelheim Investigational Site, Badalona / Barcelona
  - 135.312.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 135.312.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 135.312.34003 Boehringer Ingelheim Investigational Site, Barcelona
  - 135.312.34011 Boehringer Ingelheim Investigational Site, Bilbao
  - 135.312.34007 Boehringer Ingelheim Investigational Site, Girona
  - 135.312.34009 Boehringer Ingelheim Investigational Site, Madrid
  - 135.312.34010 Boehringer Ingelheim Investigational Site, Madrid
  - 135.312.34020 Boehringer Ingelheim Investigational Site, Madrid
  - 135.312.34017 Boehringer Ingelheim Investigational Site, Santiago de Compostela
  - 135.312.34018 Boehringer Ingelheim Investigational Site, Seville
  - 135.312.34014 Boehringer Ingelheim Investigational Site, Zaragoza
- Sweden (5):
  - 135.312.46007 Boehringer Ingelheim Investigational Site, Lidköping
  - 135.312.46003 Boehringer Ingelheim Investigational Site, Malmo
  - 135.312.46005 Boehringer Ingelheim Investigational Site, Skövde
  - 135.312.46002 Boehringer Ingelheim Investigational Site, Stockholm
  - 135.312.46004 Boehringer Ingelheim Investigational Site, Stockholm
- Switzerland (4):
  - 135.312.41003 Boehringer Ingelheim Investigational Site, Aarau
  - 135.312.41001 Boehringer Ingelheim Investigational Site, Basel
  - 135.312.41004 Boehringer Ingelheim Investigational Site, Lausanne
  - 135.312.41002 Boehringer Ingelheim Investigational Site, Sankt Gallen
- United Kingdom (9):
  - 135.312.44025 Boehringer Ingelheim Investigational Site, Aberdeen
  - 135.312.44002 Boehringer Ingelheim Investigational Site, Bournemouth
  - 135.312.44023 Boehringer Ingelheim Investigational Site, Cambridge
  - 135.312.44026 Boehringer Ingelheim Investigational Site, Dundee
  - 135.312.44003 Boehringer Ingelheim Investigational Site, Glasgow
  - 135.312.44006 Boehringer Ingelheim Investigational Site, Glasgow
  - 135.312.44024 Boehringer Ingelheim Investigational Site, Glasgow
  - 135.312.44018 Boehringer Ingelheim Investigational Site, Liverpool
  - 135.312.44030 Boehringer Ingelheim Investigational Site, London

REFERENCES:
- [Derived] Alper BS, Foster G, Thabane L, Rae-Grant A, Malone-Moses M, Manheimer E. Thrombolysis with alteplase 3-4.5 hours after acute ischaemic stroke: trial reanalysis adjusted for baseline imbalances. BMJ Evid Based Med. 2020 Oct;25(5):168-171. doi: 10.1136/bmjebm-2020-111386. Epub 2020 May 19. PMID 32430395
- [Derived] Bluhmki E, Chamorro A, Davalos A, Machnig T, Sauce C, Wahlgren N, Wardlaw J, Hacke W. Stroke treatment with alteplase given 3.0-4.5 h after onset of acute ischaemic stroke (ECASS III): additional outcomes and subgroup analysis of a randomised controlled trial. Lancet Neurol. 2009 Dec;8(12):1095-102. doi: 10.1016/S1474-4422(09)70264-9. Epub 2009 Oct 21. PMID 19850525
- [Derived] Hacke W, Kaste M, Bluhmki E, Brozman M, Davalos A, Guidetti D, Larrue V, Lees KR, Medeghri Z, Machnig T, Schneider D, von Kummer R, Wahlgren N, Toni D; ECASS Investigators. Thrombolysis with alteplase 3 to 4.5 hours after acute ischemic stroke. N Engl J Med. 2008 Sep 25;359(13):1317-29. doi: 10.1056/NEJMoa0804656. PMID 18815396